CLINICAL TRIAL: NCT00003777
Title: A Pilot Study of Combined Modality Therapy for Recurrent Head and Neck Carcinoma
Brief Title: Surgery, Radiation Therapy, and Combination Chemotherapy in Treating Patients With Recurrent Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Purpose: Treatment
Other Study IDs: CDR0000066906; UPCC-6398; ALZA-98-023-ii; NCI-V99-1518
Record Dates: First submitted 1999-11-01; First posted 2003-12-10 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent laryngeal cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Amifostine; Cisplatin; Fluorouracil; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: fluorouracil
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as amifostine may prevent the side effects of radiation therapy. Combining more than one drug and combining radiation therapy and surgery with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining surgery, radiation therapy, and combination chemotherapy in treating patients who have recurrent head and neck cancer that has been treated previously with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness and toxic effects of intensive salvage therapy and radiotherapy in previously irradiated patients with recurrent head and neck cancer.
* Determine the feasibility and effectiveness of amifostine at limiting or minimizing side effects of repeat irradiation in these patients.

OUTLINE: Patients undergo surgical resection of gross disease (if not already done) followed by 4-6 weeks of rest. Patients receive radiotherapy over 5 consecutive days on weeks 1, 2, 4, and 5. Intravenous cisplatin is administered on days 1-3 and 29-31. Intravenous amifostine is administered 15-30 minutes prior to radiotherapy and cisplatin therapy. Patients receive fluorouracil IV continuously on days 1-4 and 29-32.

Patients are followed every month for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or new primary squamous cell carcinoma of the head and neck occurring in a previously irradiated field
* Pathologic stage of recurrence must be rT3-4 and/or rN2-3
* The following sites are eligible:

  * Oral cavity, oropharynx, or hypopharynx: Any rT2-4 and/or clinical rN+
  * Larynx: Any rT4, rT3 with perineural invasion, or any rT with clinical rN+
  * Any site: Positive margin(s), at least 2 nodes or ECS
* No primary tumor of the nasopharynx
* Must be eligible for or have undergone complete resection which leaves behind no gross residual disease
* Must have prior head and neck irradiation of 45-75 Gy
* Lifetime spinal cord radiotherapy dose no greater than 50 Gy
* No ongoing RTOG late morbidity of grade 3 or greater (unless correctable by surgery)
* No active acute radiation mucositis from previous radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT or SGPT no greater than 3 times upper limit of normal
* Bilirubin no greater than 2 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No myocardial infarction, unstable angina, coronary heart failure, or uncontrolled arrhythmias within past 6 months
* No severe cerebrovascular disease or hypotension not caused by antihypertensive medication

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No allergy to cisplatin, fluorouracil, or amifostine
* No uncontrolled insulin-dependent diabetes mellitus or other medical condition interfering with wound healing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for tumor recurrence (except adjuvant chemotherapy)

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 6 months since prior radiotherapy
* Prior radiotherapy treatment records must be available

Surgery:

* No prior salvage surgery consisting of partial laryngectomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1998-12 (Actual); Primary Completion 2001-04 (Actual); Study Completion 2001-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania, United States